CLINICAL TRIAL: NCT04070937
Title: Correlation of Radiological Lesions With Vestibular Function in Patients With Bilateral Vestibulopathy
Status: Recruiting | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Sebastien Janssens de Varebeke, principal investigator, Jessa Hospital
Other Study IDs: JessaH-4
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hearing Loss, Sensorineural; Bilateral Vestibular Deficiency; DFNA9; Radiology
MeSH Terms: conditions — Hearing Loss, Sensorineural; Bilateral Vestibulopathy | interventions — Vestibular Evoked Myogenic Potentials; Audiometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — from all patients presenting bilateral vestibulopathy samples will be taken to investigate presence of p.P51S mutation in COCH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: all patients at least 18 years of age who present bilateral vestibulopathy on vestibular investigations according to the Barany criteria
  Interventions: Diagnostic Test: vestibular test 1; Diagnostic Test: vestibular test 2; Diagnostic Test: vestibular evoked myogenic potentials; Diagnostic Test: audiometry; Diagnostic Test: CT and MR imaging of temporal bone; Genetic: p.P51S mutation
- control group: DFNA9 patients carrying the p.P51S mutation in COCH gene presenting bilateral vestibulopathy according to the Barany criteria
  Interventions: Diagnostic Test: vestibular test 1; Diagnostic Test: vestibular test 2; Diagnostic Test: vestibular evoked myogenic potentials; Diagnostic Test: audiometry; Diagnostic Test: CT and MR imaging of temporal bone; Genetic: p.P51S mutation

INTERVENTIONS:
Diagnostic Test: vestibular test 1 — videonystagmography
Diagnostic Test: vestibular test 2 — video head impulse test
Diagnostic Test: vestibular evoked myogenic potentials — vestibular evoked myogenic potentials to measure the function of otolith organs
Diagnostic Test: audiometry — tonal liminar audiometric thresholds
Diagnostic Test: CT and MR imaging of temporal bone — Ct and MR imaging of temporal bone
Genetic: p.P51S mutation — analysis of presence of p.P51S mutation in COCH

SUMMARY:
In 2014 radiologic lesions were detected at one or more semicircular canals using CT and MR imaging of temporal bone in subjects carrying the p.P51S mutation in COCH. These lesions are believed to present at more advanced stages of the hearing and vestibular deterioration. Since then, other authors have described similar lesions in advanced non-genetic hearing and vestibular impairment as well.

The purpose of this study is therefore to assess the radiologic investigation using CT and MR imaging of temporal bone to all subjects presenting with bilateral vestibulopathy, using the Barany criteria, compared to the p.P51S population.

ELIGIBILITY:
Inclusion Criteria:

* must meet the Barany criteria for bilateral vestibulopathy: bilaterally pathological horizontal angu- lar VOR gain <0.6, measured by the video-HIT5 or scleral-coil technique and/or
* reduced caloric response6 (sum of bither- mal max. peak SPV on each side <6◦/sec7) and/or
* reduced horizontal angular VOR gain <0.1 upon sinusoidal stimulation on a rota- tory chair (0.1 Hz, Vmax = 50◦ /sec) and a phase lead >68 degrees (time constant <5 sec).
* must be 18 or older

Exclusion Criteria:

* < 18 y
* does not meet Barany criteria for BV
* contraindication for CT and MR imaging

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients presenting at our Department of ENT with vestibular or balance disorders, in whom videonystagmography, video head impulse test and VEMP tests meet the Barany criteria for bilateral vestibulopathy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
CT and MR findings | at time of recruitment
  presence of focal sclerosis or signal loss on CT & MR at one or more semicircular canals
genetic test | at time of recruitment
  p.P51S mutation in COCH gene

SECONDARY OUTCOMES:
vestibular test 1 | at time of recruitment
  video nystagmography using caloric tests ; caloric tests: °/s
vestibular test 2 | at time of recruitment
  video head impulse test; gain for each SCC in °/s
vestibular test 3 | at time of recruitment
  vestibular evoked myogenic potentials: threshold in decibel normal hearing loss (dB nHL)
audiometry | at time of recruitment
  tonal liminar audiometry using calibrated audiometer, threshold in dB HL

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No